CLINICAL TRIAL: NCT02442102
Title: Understanding and Improving Dysphagia After Mechanical Ventilation
Brief Title: PReventing the EffectS of Intubation on DEglutition
Acronym: PRESIDE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow recruitment
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00029289; 1K23DC013569-01 (NIH)
Record Dates: First submitted 2015-05-04; First posted 2015-05-13 (Estimated); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Deglutition Disorders; Mechanical Ventilation Complication; Complication of Ventilation Therapy
Keywords: deglutition disorders; therapeutics; rehabilitation; outcome assessment; intubation; critical care; larynx; voice
MeSH Terms: conditions — Deglutition Disorders; Laryngeal Diseases | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise and sensory stimulation (Experimental): 60-minute sessions with sensory electrical stimulation (SES) applied 5 days per week with oromotor exercises completed when patient is able to participate
  Interventions: Behavioral: Exercise and sensory stimulation

INTERVENTIONS:
Behavioral: Exercise and sensory stimulation — 60-minute sessions with sensory electrical stimulation (SES) applied 5 days per week with oromotor exercises completed when patient is able to participate
  Other Names: VitalStim (Chattanooga Group; Hixson, TN)

SUMMARY:
An early intervention for swallowing disorders (i.e., dysphagia) during endotracheal intubation may improve patient outcomes. The investigators propose treatment sessions targeting sensorimotor integration, strength, and range of motion during oral endotracheal intubation with mechanical ventilation to reduce or prevent dysphagia and aspiration (food or liquids entering the airway), establish a solid foundation in understanding reasons for swallowing impairment after extubation from mechanical ventilation and learn new methods to reduce or prevent these problems.

DETAILED DESCRIPTION:
The overall goals of this study are to evaluate patients with acute respiratory failure from the time they are orally intubated in the ICU to: 1) investigate tongue weakness and other pathophysiological aspects of dysphagia, and 2) evaluate, in a Phase II clinical trial, a novel, multimodal, sensorimotor intervention conducted during intubation to reduce or prevent dysphagia after extubation. Patients who are expected to be intubated with mechanical ventilation for >96 hours will be consecutively enrolled shortly after intubation. Laryngeal function, tongue strength, swallowing pathophysiology, and breathing-swallowing coordination will be evaluated with valid and reliable standardized measures. While orally intubated, patients in the treatment group will receive a novel, early, sensorimotor intervention for 60-minutes daily, 5 times per week, targeting improved swallowing physiology and kinematics to reduce aspiration and dysphagia. These daily sessions will continue until the completion of a modified barium swallow study conducted within approximately 2 days after extubation, and thereafter standard clinical care will resume. Patients in the control group will receive standard clinical care during intubation and throughout their hospital stay. All patients will be followed to hospital discharge to determine the pathophysiological and clinical impact of the proposed intervention. Knowledge from this study will provide important data for this novel intervention and provide a critical foundation for understanding the physiological mechanisms of dysphagia and aspiration after intubation in patients with acute respiratory failure. With success, this investigation will help shift clinical practice patterns to consider early intervention with the goal of reducing the frequency and severity of swallowing impairment leading to aspiration and additional medical complications.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Required mechanical ventilation via an oral endotracheal tube

Exclusion Criteria:

* Unable to understand or speak English due to a language barrier
* Unable to understand or speak English due to a cognitive impairment
* Barium sulfate allergy
* Pregnancy
* Presence of any cardiac pacing device (including temporary epicardial pacing) without an underlying cardiac rhythm as confirmed by treating physician or diaphragmatic pacer
* Nasal endotracheal intubation during the present admission
* Patient is not expected to require ≥48 hours of intubation
* Pre-existing dysphagia/aspiration, voice or cognitive disorder
* Reflux with history of known or suspected aspiration
* Presence of a central nervous system, neuromuscular or connective tissue disease (e.g., stroke, Guillain-Barre, scleroderma)
* Active seizure disorder
* Pain disorder of the jaw muscles or mandibular joint
* Ever tracheotomy or prior endotracheal intubation other than for surgery (≤ 1 year)
* Head and/or neck disease (e.g., oropharyngeal cancer)
* Head and/or neck surgery other than tonsillectomy
* Known or suspected anatomical abnormalities or pre-intubation trauma of the oral cavity, pharynx, larynx, or esophagus
* Known or suspected sleep apnea (treated or untreated)
* Prior major thoracic surgery (e.g., sternotomy, thoracotomy)
* Unplanned (e.g., self- or accidental) extubation or re-intubation before consent
* Weight exceeds capacity of the radiology equipment
* Expected tracheostomy tube placement while in hospital
* Moribund (>90% probability of mortality in hospital), based on ICU team's assessment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-07; Primary Completion 2022-08 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
Number of participants aspirating during fiberoptic endoscopic swallow study | participants will be evaluated an expected average of 48 hours after extubation

CONTACTS AND LOCATIONS:
Overall Officials: Dale M Needham, MD PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Adhikari NK, Fowler RA, Bhagwanjee S, Rubenfeld GD. Critical care and the global burden of critical illness in adults. Lancet. 2010 Oct 16;376(9749):1339-46. doi: 10.1016/S0140-6736(10)60446-1. Epub 2010 Oct 11. PMID 20934212
- [Background] Ajemian MS, Nirmul GB, Anderson MT, Zirlen DM, Kwasnik EM. Routine fiberoptic endoscopic evaluation of swallowing following prolonged intubation: implications for management. Arch Surg. 2001 Apr;136(4):434-7. doi: 10.1001/archsurg.136.4.434. PMID 11296115
- [Background] Bailey P, Thomsen GE, Spuhler VJ, Blair R, Jewkes J, Bezdjian L, Veale K, Rodriquez L, Hopkins RO. Early activity is feasible and safe in respiratory failure patients. Crit Care Med. 2007 Jan;35(1):139-45. doi: 10.1097/01.CCM.0000251130.69568.87. PMID 17133183
- [Background] Barquist E, Brown M, Cohn S, Lundy D, Jackowski J. Postextubation fiberoptic endoscopic evaluation of swallowing after prolonged endotracheal intubation: a randomized, prospective trial. Crit Care Med. 2001 Sep;29(9):1710-3. doi: 10.1097/00003246-200109000-00009. PMID 11546969
- [Background] Colice GL, Stukel TA, Dain B. Laryngeal complications of prolonged intubation. Chest. 1989 Oct;96(4):877-84. doi: 10.1378/chest.96.4.877. PMID 2791687
- [Background] Connor NP, Russell JA, Wang H, Jackson MA, Mann L, Kluender K. Effect of tongue exercise on protrusive force and muscle fiber area in aging rats. J Speech Lang Hear Res. 2009 Jun;52(3):732-44. doi: 10.1044/1092-4388(2008/08-0105). Epub 2008 Aug 22. PMID 18723593
- [Background] De Jonghe B, Cook D, Sharshar T, Lefaucheur JP, Carlet J, Outin H. Acquired neuromuscular disorders in critically ill patients: a systematic review. Groupe de Reflexion et d'Etude sur les Neuromyopathies En Reanimation. Intensive Care Med. 1998 Dec;24(12):1242-50. doi: 10.1007/s001340050757. PMID 9885875
- [Background] de Larminat V, Montravers P, Dureuil B, Desmonts JM. Alteration in swallowing reflex after extubation in intensive care unit patients. Crit Care Med. 1995 Mar;23(3):486-90. doi: 10.1097/00003246-199503000-00012. PMID 7874899
- [Background] El Solh A, Okada M, Bhat A, Pietrantoni C. Swallowing disorders post orotracheal intubation in the elderly. Intensive Care Med. 2003 Sep;29(9):1451-5. doi: 10.1007/s00134-003-1870-4. Epub 2003 Aug 2. PMID 12904855
- [Background] Hedden M, Ersoz CJ, Donnelly WH, Safar P. Laryngotracheal damage after prolonged use of orotracheal tubes in adults. JAMA. 1969 Jan 27;207(4):703-8. No abstract available. PMID 5818186
- [Background] Herridge MS, Cheung AM, Tansey CM, Matte-Martyn A, Diaz-Granados N, Al-Saidi F, Cooper AB, Guest CB, Mazer CD, Mehta S, Stewart TE, Barr A, Cook D, Slutsky AS; Canadian Critical Care Trials Group. One-year outcomes in survivors of the acute respiratory distress syndrome. N Engl J Med. 2003 Feb 20;348(8):683-93. doi: 10.1056/NEJMoa022450. PMID 12594312
- [Background] Hussain SN, Mofarrahi M, Sigala I, Kim HC, Vassilakopoulos T, Maltais F, Bellenis I, Chaturvedi R, Gottfried SB, Metrakos P, Danialou G, Matecki S, Jaber S, Petrof BJ, Goldberg P. Mechanical ventilation-induced diaphragm disuse in humans triggers autophagy. Am J Respir Crit Care Med. 2010 Dec 1;182(11):1377-86. doi: 10.1164/rccm.201002-0234OC. Epub 2010 Jul 16. PMID 20639440
- [Background] Hwang CH, Choi KH, Ko YS, Leem CM. Pre-emptive swallowing stimulation in long-term intubated patients. Clin Rehabil. 2007 Jan;21(1):41-6. doi: 10.1177/0269215506071286. PMID 17213240
- [Background] Jaber S, Petrof BJ, Jung B, Chanques G, Berthet JP, Rabuel C, Bouyabrine H, Courouble P, Koechlin-Ramonatxo C, Sebbane M, Similowski T, Scheuermann V, Mebazaa A, Capdevila X, Mornet D, Mercier J, Lacampagne A, Philips A, Matecki S. Rapidly progressive diaphragmatic weakness and injury during mechanical ventilation in humans. Am J Respir Crit Care Med. 2011 Feb 1;183(3):364-71. doi: 10.1164/rccm.201004-0670OC. Epub 2010 Sep 2. PMID 20813887
- [Background] Langmore SE, Terpenning MS, Schork A, Chen Y, Murray JT, Lopatin D, Loesche WJ. Predictors of aspiration pneumonia: how important is dysphagia? Dysphagia. 1998 Spring;13(2):69-81. doi: 10.1007/PL00009559. PMID 9513300
- [Background] Levine S, Nguyen T, Taylor N, Friscia ME, Budak MT, Rothenberg P, Zhu J, Sachdeva R, Sonnad S, Kaiser LR, Rubinstein NA, Powers SK, Shrager JB. Rapid disuse atrophy of diaphragm fibers in mechanically ventilated humans. N Engl J Med. 2008 Mar 27;358(13):1327-35. doi: 10.1056/NEJMoa070447. PMID 18367735
- [Background] Marik PE, Kaplan D. Aspiration pneumonia and dysphagia in the elderly. Chest. 2003 Jul;124(1):328-36. doi: 10.1378/chest.124.1.328. PMID 12853541
- [Background] Martin BJ, Corlew MM, Wood H, Olson D, Golopol LA, Wingo M, Kirmani N. The association of swallowing dysfunction and aspiration pneumonia. Dysphagia. 1994 Winter;9(1):1-6. doi: 10.1007/BF00262751. PMID 8131418
- [Background] Morris PE, Goad A, Thompson C, Taylor K, Harry B, Passmore L, Ross A, Anderson L, Baker S, Sanchez M, Penley L, Howard A, Dixon L, Leach S, Small R, Hite RD, Haponik E. Early intensive care unit mobility therapy in the treatment of acute respiratory failure. Crit Care Med. 2008 Aug;36(8):2238-43. doi: 10.1097/CCM.0b013e318180b90e. PMID 18596631
- [Background] Needham DM. Mobilizing patients in the intensive care unit: improving neuromuscular weakness and physical function. JAMA. 2008 Oct 8;300(14):1685-90. doi: 10.1001/jama.300.14.1685. PMID 18840842
- [Background] Needham DM, Korupolu R, Zanni JM, Pradhan P, Colantuoni E, Palmer JB, Brower RG, Fan E. Early physical medicine and rehabilitation for patients with acute respiratory failure: a quality improvement project. Arch Phys Med Rehabil. 2010 Apr;91(4):536-42. doi: 10.1016/j.apmr.2010.01.002. PMID 20382284
- [Background] Orlikowski D, Terzi N, Blumen M, Sharshar T, Raphael JC, Annane D, Lofaso F. Tongue weakness is associated with respiratory failure in patients with severe Guillain-Barre syndrome. Acta Neurol Scand. 2009 Jun;119(6):364-70. doi: 10.1111/j.1600-0404.2008.01107.x. Epub 2008 Oct 22. PMID 18976323
- [Background] Robbins J, Gangnon RE, Theis SM, Kays SA, Hewitt AL, Hind JA. The effects of lingual exercise on swallowing in older adults. J Am Geriatr Soc. 2005 Sep;53(9):1483-9. doi: 10.1111/j.1532-5415.2005.53467.x. PMID 16137276
- [Background] Robbins J, Kays SA, Gangnon RE, Hind JA, Hewitt AL, Gentry LR, Taylor AJ. The effects of lingual exercise in stroke patients with dysphagia. Arch Phys Med Rehabil. 2007 Feb;88(2):150-8. doi: 10.1016/j.apmr.2006.11.002. PMID 17270511
- [Background] Schweickert WD, Hall J. ICU-acquired weakness. Chest. 2007 May;131(5):1541-9. doi: 10.1378/chest.06-2065. PMID 17494803
- [Background] Schweickert WD, Pohlman MC, Pohlman AS, Nigos C, Pawlik AJ, Esbrook CL, Spears L, Miller M, Franczyk M, Deprizio D, Schmidt GA, Bowman A, Barr R, McCallister KE, Hall JB, Kress JP. Early physical and occupational therapy in mechanically ventilated, critically ill patients: a randomised controlled trial. Lancet. 2009 May 30;373(9678):1874-82. doi: 10.1016/S0140-6736(09)60658-9. Epub 2009 May 14. PMID 19446324
- [Background] Sharshar T, Ross ET, Hopkinson NS, Porcher R, Nickol AH, Jonville S, Dayer MJ, Hart N, Moxham J, Lofaso F, Polkey MI. Depression of diaphragm motor cortex excitability during mechanical ventilation. J Appl Physiol (1985). 2004 Jul;97(1):3-10. doi: 10.1152/japplphysiol.01099.2003. Epub 2004 Mar 12. PMID 15020575
- [Background] Whited RE. A prospective study of laryngotracheal sequelae in long-term intubation. Laryngoscope. 1984 Mar;94(3):367-77. doi: 10.1288/00005537-198403000-00014. PMID 6700353
- [Background] Wunsch H, Linde-Zwirble WT, Angus DC, Hartman ME, Milbrandt EB, Kahn JM. The epidemiology of mechanical ventilation use in the United States. Crit Care Med. 2010 Oct;38(10):1947-53. doi: 10.1097/CCM.0b013e3181ef4460. PMID 20639743
- [Background] Yeates EM, Molfenter SM, Steele CM. Improvements in tongue strength and pressure-generation precision following a tongue-pressure training protocol in older individuals with dysphagia: three case reports. Clin Interv Aging. 2008;3(4):735-47. doi: 10.2147/cia.s3825. PMID 19281066